CLINICAL TRIAL: NCT04125420
Title: Hypersensitivity Reactions During Anesthesia: A Single Center Study
Brief Title: Hypersensitivity Reactions During Anesthesia
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexei Gonzalez-Estrada, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 18-001390
Record Dates: First submitted 2019-07-28; First posted 2019-10-14 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers are trying to study the natural history of allergic reactions during anesthesia and its causes and risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients over age 18 undergoing surgery at Mayo Clinic Florida

Exclusion Criteria:

* Minors under age 18
* Unable to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults undergoing surgery at Mayo Clinic Florida
Sampling Method: Non-Probability Sample
Enrollment: 940 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence. | 2-3 years
  Current estimates are between 1:400 to 1:10,000 surgeries mostly based on retrospective reviews. We will report incidence based on numbers of event/number of surgeries

SECONDARY OUTCOMES:
Risk factors | 2-3 years
  Risk factors; including female gender, prior reactions during surgery, sensitization to a previous agent used during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Gonzalez Estrada, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials